CLINICAL TRIAL: NCT01222182
Title: Statin Therapeutic Interchange by Pharmacist Collaborative Practice Process
Brief Title: Statin Interchange by Pharmacist Collaborative Practice Agreement (CPA)
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Robert Hoel, PharmD, RPh, Mayo Clinic
Other Study IDs: 10-000986
Record Dates: First submitted 2010-09-24; First posted 2010-10-18 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: Hypercholesterolemia
Keywords: low density lipoprotein (LDL) cholesterol; statin; dose equivalent; Hypercholesterolemia (defined by LDL guidelines)
MeSH Terms: conditions — Hypercholesterolemia | interventions — Atorvastatin; Pravastatin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Eligible plan beneficiaries on atorvastatin: A group of 225 eligible patients would no longer have atorvastatin covered by their prescription plan and would need to be changed to another equivalent anti-hyperlipidemic agent.
  Interventions: Drug: atorvastatin

INTERVENTIONS:
Drug: atorvastatin — All patients desired to change atorvastatin 10, 20mg to an equivalent that is covered by their prescription plan. This is accomplished by either pharmacists by MD/Pharmacist practice agreement or physicians in usual practice
  Other Names: atorvastatin, (Lipitor®),; interchanged to simvastatin, pravastatin

SUMMARY:
A group of ~ 225 patients were switched from atorvastatin to an equivalent statin either by their physicians usual management or by an collaborative pharmacist coordinated process. We will compare the results of pharmacist process to the standard medical practice to find potentially which process is more effective, safer and efficient. We are surveying a total of 35 physicians, 12 using the pharmacist coordinated process and 23 not, comparing their satisfaction of the 2 processes.

DETAILED DESCRIPTION:
This study is a retrospective analysis of patients converted from atorvastatin to another equivalent statin. It is observational because the patients were all on atorvastatin, had been informed by their prescription drug plan that it would not be covered, and that if agreed they would be changed to an equivalent that is covered by their plan. The patients were either converted with the help of pharmacist by collaborative practice agreement (CPA)or upon contacting their physician requesting a different medication. We are comparing the percentage first converted to the equivalent dose in each group and whether patients continued to be at hyperlipidemia treatment goal after the interchange.

ELIGIBILITY:
225 insured eligible subjects, 35 PCIM physicians

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 225 insured eligible subjects, 35 Primary Care Internal Medicine (PCIM) physicians
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2009-09; Primary Completion 2011-02 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Determine if a process of pharmacist practice agreement is effective in changing from atorvastatin 10, 20mg to a therapeutic equivalent dose. | 3 to 9 months after conversion from atorvastatin
  We compared doses selected for therapeutic equivalency for the new statin Did the process result in selecting a safe and effective statin alternative?

SECONDARY OUTCOMES:
Was the process regarded as efficient and satisfying to physician compared to usual practice. | 5 months post conversion
  A satisfaction survey of physicians who utilized the pharmacist collaborative practice agreement(CPA) will be compared to satisfaction of phycians who were not able to use the CPA. Was the process regarded as efficient and satisfying to physician compared to usual practice.
Did the patients' low density lipoprotein(LDL) cholesterol require further statin dose intervention? | 6-12 months
  Of patients who had a follow up LDL cholesterol, how many required another intervention after failing to stay within treatment goal. Physicians usually measure each of these patients within 3 months of a change of treatment and annually thereafter. We will look at follow up LDL cholesterol and liver function test (LFT) as recommended.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Odell, PharmD, RPh, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States